CLINICAL TRIAL: NCT05691244
Title: A Multicentric, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Study to Assess the Safety and Efficacy of Sovateltide in Patients With Acute Cerebral Ischemic Stroke.
Brief Title: Assess the Safety and Efficacy of Sovateltide in Patients With Acute Cerebral Ischemic Stroke
Acronym: RESPECT-ETB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sovateltide/ACIS/IND2022
Record Dates: First submitted 2023-01-11; First posted 2023-01-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke; Cerebral Stroke
Keywords: Endothelin B Receptors
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Saline Solution; sovateltide

STUDY DESIGN:
Intervention Model Description: This is a multi-centric, randomized, double-blind, placebo-controlled phase-III clinical study to assess the safety and efficacy of sovateltide in patients with acute cerebral ischemic stroke.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, the subject and all relevant personnel involved with the conduct and interpretation of the study (including investigator, investigational site personnel, and the sponsor or designee's staff) will remain blinded to the identity of the Investigational Product (IP) assigned and the randomization codes. The final randomization list will be kept strictly confidential, filed securely by the independent biostatistician, and accessible only to authorized persons as per the sponsor's standard operating procedures until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Saline + Standard of care (Active Comparator): Normal saline will be used as a comparator. It will be available in a 5.0 mL vial. Three doses will be administered as an IV bolus over one minute every 3 hours ± 1 hour on day 1. The dose will be repeated on days 3 and 6 post randomization. The study drug will be administered as an IV bolus dose over 1 minute within 24 hours of the stroke onset.
  Interventions: Drug: Drug: Normal Saline
- Sovateltide + Standard of care (Experimental): The test product is sovateltide. It is available as a lyophilized injection containing 30 µg of sovateltide in a 5.0 mL vial. Three doses of 0.3 μg/kg will be administered as an IV bolus over one minute every 3 hours ± 1 hour on day 1. The dose will be repeated on days 3 and 6 post randomization. The study drug will be administered as an IV bolus dose over 1 minute within 24 hours of the stroke onset.
  Interventions: Drug: Sovateltide

INTERVENTIONS:
Drug: Drug: Normal Saline — Normal saline to be used as vehicle in the phase-III study to assess efficacy of sovateltide in patients with acute cerebral ischemic stroke.
  Other Names: Vehicle
  Arms: Normal Saline + Standard of care
Drug: Sovateltide — Phase-III study to assess efficacy of sovateltide in patients with acute cerebral ischemic stroke.
  Other Names: PMZ-1620
  Arms: Sovateltide + Standard of care

SUMMARY:
Extensive research is being conducted in search of neuroprotective agents for possible use in the acute phase of stroke and agents that can be used for neurorepair in later stages of stroke. Several trials have been conducted and are in progress using different pharmacological agents, but none of the studies involve the stimulation of ETB receptors to treat cerebral ischemic stroke. Sovateltide (IRL-1620, PMZ-1620) has been effective in animal models of cerebral ischemic stroke. Its safety and tolerability have been demonstrated in a human phase I study with 7 subjects. Clinical phase II and III results indicate that sovateltide is a novel, first-in-class, highly effective drug candidate for treating cerebral ischemic stroke. Safety and significant efficacy in improving the National Institutes of Health Stroke Scale (NIHSS), Modified Rankin scale (mRS), and Barthel index (BI) obtained in phase II and III studies in patients with cerebral ischemic stroke in India are convincing and encouraged us to investigate its safety and efficacy in cerebral ischemic stroke patients in the United States. Therefore, the plan is to conduct a phase III clinical study to evaluate the safety and efficacy of sovateltide therapy along with standard of care in patients of acute ischemic stroke.

DETAILED DESCRIPTION:
A stroke is a syndrome defined as an abrupt neurological outburst due to impaired blood flow to part of the brain. There are two types of stroke: hemorrhagic stroke and ischemic stroke. A hemorrhagic stroke follows the rupture of a weakened blood vessel in the brain causing accumulation of blood and compression of the surrounding brain tissue. An ischemic stroke follows a blocked blood vessel by a thrombus (blood clot) or embolism. In both types of strokes, the specific region of the brain supplied by the affected blood vessel is deprived of oxygenated blood, causing local hypoxia that damages the brain tissue and cells. Both types of stroke are very serious, however ischemic stroke is more common.

The global burden of ischemic stroke is nearly 4-fold greater than hemorrhagic stroke with close to 87% of the total incidence of stroke attributed to acute cerebral ischemic stroke (ACIS). ACIS is a critical care emergency caused by a significant reduction in blood flow to the brain by a blood clot or embolism. This nearly halts cerebral blood flow to the affected region leading to neuronal death. Neuronal cell death is followed by plasma membrane disruption, swelling of organelles, leaking of cell contents into extracellular space, and loss of neuronal function. Other events that take place include inflammation, excitotoxicity, free radical mediated toxicity, cytokine mediated cytotoxicity, impaired blood-brain-barrier, and oxidative stress.

Therapeutic management of ACIS is a multidisciplinary approach with a primary goal of revascularization and limiting neuronal injury. A stroke team consists of emergency medicine physicians, neurologists/neurosurgeons, radiologists, nurses and advanced care providers, clinical pharmacists, therapists, technicians, and laboratory personnel. Currently, the only FDA-approved pharmacological agent for ischemic stroke is tissue plasminogen activator (t-PA). It is a thrombolytic agent which restores blood flow by breaking down a clot. However, timing is crucial in administration of t-PA as the therapeutic time window is very narrow and the patient must receive it within 4.5 hours of onset of stroke symptoms. Therapeutic administration after this timeframe can result in hemorrhagic transformation, leading to additional brain damage. Nevertheless, even upon timely administration of t-PA in ACIS, only about 30% of patients obtain stroke resolution having minimal or no disability at the 90-day mark.

Sovateltide (PMZ-1620, IRL-1620) is a highly selective ETB receptor agonist and a synthetic analog of ET-1. Studies conducted to determine the effects brought about by sovateltide upon its interaction with neural ETB receptors and have found that it enhances angiogenesis and neurogenesis as well as promotes neural repair and regeneration. In a rat model of ischemic stroke, sovateltide was found to be neuroprotective as well as enhance angiogenic and neurogenic remodeling. Sovateltide significantly improved survival, reduced neurological and motor function deficit, while effectively decreasing infarct volume, edema, and oxidative stress.

Sovateltide was also found to be safe and well tolerated in healthy human volunteers in a phase I clinical trial (CTRI/2016/11/007509). A phase II study was also conducted in patients with acute ischemic stroke where sovateltide demonstrated significant improvement when compared to standard of care (CTRI/2017/11/010654, NCT04046484). A recent phase III study conducted in patients of acute ischemic stroke demonstrated improved favorable functional and neurological outcome at 3 months compared to standard of care (CTRI/2019/09/021373, NCT04047563).

Clinical phase II and III results indicate that sovateltide is a first-in-class neuronal progenitor cell therapeutic that promotes quick recovery and significantly improves neurological outcomes in cerebral ischemic stroke patients. With this convincing evidence, the plan is to conduct a multicentric, randomized, double-blind, parallel, placebo-controlled phase III clinical study in the United States, Canada, United Kingdom and Europe (the demographics and standard of treatment being similar in these countries) to further assess the safety and efficacy of sovateltide in patients with acute cerebral ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in the study if he/she fulfills the following criteria:

1. Adult males or females aged 18 - 80 years of age.
2. Consent obtained per national laws and regulations, and in accordance with the applicable ethics committee requirements prior to study procedures.
3. A stroke is ischemic in origin that is diagnosed clinically and/or radiologically confirmed by Computed Tomography (CT) scan or diagnostic magnetic resonance imaging (MRI) prior to enrolment. No hemorrhage as proved by cerebral CT/MRI scan.
4. Cerebral ischemic stroke patients presenting within 24 hours after the onset of symptoms with NIHSS score of ≥8 and <20, NIHSS Level of Consciousness (1A) score <2 at the time of screening. This includes cerebral ischemic stroke patients who completely recovered from earlier episodes before having a new or fresh stroke having a pre-stroke historical measure of mRS score of 0-2.
5. The patient is <24 hours from the time of stroke onset when the first dose of sovateltide is administered. Time of onset is when symptoms began; for stroke that occurred during sleep, time of onset is when the patient was last seen or was self- reported to be normal.
6. Reasonable expectation of availability to receive the full sovateltide/placebo course of therapy and to be available for subsequent follow-up visits.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if they meet any of the following exclusion criteria:

1. Patients receiving endovascular therapy or is a candidate for any surgical intervention for the treatment of stroke, which may include but not limited to endovascular techniques.
2. Patients classified as comatose are defined as a patient who requires repeated stimulation to attend or is obtunded and requires strong or painful stimulation to make movements (NIHSS Level of Consciousness (1A) score ≥2).
3. Evidence of intracranial hemorrhage (intracerebral hematoma, intraventricular hemorrhage, subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on the baseline CT or MRI scan.
4. Known pregnancy and lactating women.
5. Known medical history of neurological (other than current acute ischemic stroke) or psychiatric condition that, in the investigator's opinion, would confound the neurological and functional evaluations, lead to further deterioration of neurological status, or interfere with participation in this study.
6. Concurrent participation in any other therapeutic clinical trial.
7. Evidence of any other major life-threatening or serious medical condition that would prevent completion of the study protocol impair the assessment of outcome, or in which sovateltide therapy would be contraindicated or might cause harm to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of sovateltide in patients with acute cerebral ischemic stroke assessed by modified Rankin Scale (mRS) score of 0-2 at day 90 post-randomization. | Day 1 through Day 90
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with a modified Rankin Scale score of 0-2 on day 90 post-randomization.

SECONDARY OUTCOMES:
Determine a good functional outcome in patients with acute cerebral ischemic stroke assessed by the National Institute of Health Stroke Scale (NIHSS) score of <6 at day 90 post-randomization. | Day 1 through Day 90
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with NIHSS score of <6 on day 90 post-randomization.
Determine a good functional outcome in patients with acute cerebral ischemic stroke assessed by the Barthel Index (BI) score of ≥90 at day 90 post-randomization. | Day 1 through Day 90
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with BI score of ≥90 on day 90 post-randomization.
Determine an excellent functional outcome in patients with acute cerebral ischemic stroke assessed by a modified Rankin Scale score of 0-1 at day 90 post-randomization. | Day 1 through Day 90
  The proportion of acute cerebral ischemic stroke patients having an excellent functional outcome with a modified Rankin Scale score of 0-1 on day 90 post-randomization.
Determine a change in Quality-of-life (QoL) as assessed by EuroQol-EQ-5D-5L and Stroke-Specific Quality of Life (SS-QOL) at days 30, 60, and 90 post-randomization. | Day 1 through Day 90
  Change in QoL as assessed by EuroQol EQ-5D-5L and by SS-QOL from baseline to days 30, 60, and 90 post-randomization.
Determine the incidence of recurrent cerebral ischemic stroke within 90 days post-randomization. | Day 1 through Day 90
  The proportion of patients with recurrent ischemic stroke within 90 days post-randomization.
Determine the incidence of mortality within 90 days post-randomization. | Day 1 through Day 90
  Number of deaths within day 90 post-randomization.
Determine the incidence of symptomatic Intracerebral Hemorrhage (ICH) within 24 (± 6) hours of randomization. | Day 1 through Day 90
  The proportion of patients with symptomatic ICH within 24 (± 6) hours of randomization.
Determine the incidence of radiographic Intracerebral Hemorrhage (ICH) within 24 (± 6) hours of randomization. | Day 1 through Day 90
  The proportion of patients with radiographic ICH within 24 (± 6) hours of randomization.
Determine alteration in cognition at days 30 and 90 measured by Montreal Cognitive Assessment (MoCA) Test. | Day 1 through Day 90
  Change in MoCA score at days 30 and 90 post-randomization.
Determine any adverse events (AE) or serious adverse events (SAEs) are associated with sovateltide. | Day 1 through Day 90
  The proportion of patients with adverse events (AEs) and serious adverse events (SAEs).

OTHER OUTCOMES:
Determine a good functional outcome in patients with acute cerebral ischemic stroke assessed by mRS score of 0-2 at day 30 post-randomization. | Day 1 through Day 30
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with a mRS score of 0-2 on day 30 post-randomization.
Determine a good functional outcome in patients with acute cerebral ischemic stroke assessed by the NIHSS score of <6 at day 30 post-randomization. | Day 1 through Day 30
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with NIHSS score of <6 on day 30 post-randomization.
Determine a good functional outcome in patients with acute cerebral ischemic stroke assessed by the BI score of ≥90 at day 30 post-randomization. | Day 1 through Day 30
  The proportion of acute cerebral ischemic stroke patients having a good functional outcome with BI score of ≥90 on day 30 post-randomization.
Determine Alberta Stroke Program Early CT (ASPECT) Score for stroke severity at baseline and identify sites of ischemic lesions. | Day 1 through Day 90
  Compare baseline Alberta Stroke Program Early CT (ASPECT) Score for stroke severity and identify sites of ischemic lesions.
Determine the subtype of acute cerebral ischemic stroke according to TOAST classification at day 30 post-randomization. | Day 1 through Day 30
  Compare the subtype of acute cerebral ischemic stroke by TOAST classification at day 30 post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, MD, PhD, Study Chair — Pharmazz, Inc.
Locations (42):
- United States (9):
  - The University of Arizona - College of Medicine, Tuscon, Arizona
  - Mercy Medical Group, Carmichael, California
  - St. John's Regional Medical Center, Oxnard, California
  - SSM Health Neurosciences, Bridgeton, Missouri
  - OSU Wexner Medical Center, Columbus, Ohio
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - CHI Memorial Neuroscience Institute, Chattanooga, Tennessee
  - Houston Medical Neurological Institute, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
- Germany (8):
  - Klinikum Altenburger Land GmbH, Altenburg, Altenburg
  - Universitaetsklinikum Goettingen, Göttingen, Lower Saxony
  - Klinikum der Stadt Ludwigshafen gGmbh, Rhein, Ludwigshafen Am
  - Muhlenkreiskliniken (MKK) - Johannes Wesling Klinikum Minden - Neurologische Klinik, Minden, North Rhine-Westphalia
  - Klinik fuer Neurologie, Stroke Unit und Fruehrehabilitation Dorstener Strae 151, Recklinghausen, Recklinghausen
  - Charite-Universitaetsmedizin Berlin, Berlin, State of Berlin
  - Universitätsklinikum Essen AöR, Essen
  - Universitätsklinikum Schleswig-Holstein AöR, Lübeck
- Spain (19):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Complejo Hospitalario Universitario de Albacete, Albacete, Castille-La Mancha
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de Arrixaca, El Palmar, Murcia
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Joan XXIII, Tarragona, Tarragona
  - Instituto de Investigación Biomédica de A Coruña, A Coruña
  - Hospital Universitario Infanta Cristina (HUB), Badajoz
  - Hospital Universitario de Cruces, Barakaldo
  - Institut Catala d'Oncologia (ICO) - Hospital Universitari Doctor Josep Trueta, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Fairfield General Hospital, Bury, Bury
  - National Hospital for Neurology & Neurosurgery, London, London
  - King's College Hospital NHS Foundation Trust, London, London
  - University Hospital Southampton, Southampton, Southampton
  - New Cross Hospital - Royal Wolverhampton NHS Trust, Wolverhampton, Wolverhampton
  - Hospitals NHS Foundation Trust - Royal Victoria Infirmary RVI, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the trial in 2027, the anonymized patient datasets created and/or analyzed for the current study can be accessed from the corresponding author at a reasonable request from a bona fide researcher/research group.
Supporting Information: Study Protocol
Time Frame: December 2027
Access Criteria: Following completion of the trial in 2027, the anonymized patient datasets created and/or analyzed for the current study can be accessed from the corresponding author at a reasonable request from a bona fide researcher/research group.

REFERENCES:
- [Background] Gulati A, Adwani SG, Vijaya P, Agrawal NR, Ramakrishnan TCR, Rai HP, Jain D, Sundarachary NV, Pandian JD, Sardana V, Sharma M, Sidhu GK, Anand SS, Vibha D, Aralikatte S, Khurana D, Joshi D, Karadan U, Siddiqui MSI. Efficacy and Safety of Sovateltide in Patients with Acute Cerebral Ischaemic Stroke: A Randomised, Double-Blind, Placebo-Controlled, Multicentre, Phase III Clinical Trial. Drugs. 2024 Dec;84(12):1637-1650. doi: 10.1007/s40265-024-02121-5. Epub 2024 Nov 15. PMID 39542995
- [Background] Ranjan AK, Gulati A. Sovateltide Mediated Endothelin B Receptors Agonism and Curbing Neurological Disorders. Int J Mol Sci. 2022 Mar 15;23(6):3146. doi: 10.3390/ijms23063146. PMID 35328566
- [Background] Gulati A, Agrawal N, Vibha D, Misra UK, Paul B, Jain D, Pandian J, Borgohain R. Safety and Efficacy of Sovateltide (IRL-1620) in a Multicenter Randomized Controlled Clinical Trial in Patients with Acute Cerebral Ischemic Stroke. CNS Drugs. 2021 Jan;35(1):85-104. doi: 10.1007/s40263-020-00783-9. Epub 2021 Jan 11. PMID 33428177
- [Background] Ramos MD, Briyal S, Prazad P, Gulati A. Neuroprotective Effect of Sovateltide (IRL 1620, PMZ 1620) in a Neonatal Rat Model of Hypoxic-Ischemic Encephalopathy. Neuroscience. 2022 Jan 1;480:194-202. doi: 10.1016/j.neuroscience.2021.11.027. Epub 2021 Nov 23. PMID 34826534
- [Background] Ranjan AK, Briyal S, Gulati A. Sovateltide (IRL-1620) activates neuronal differentiation and prevents mitochondrial dysfunction in adult mammalian brains following stroke. Sci Rep. 2020 Jul 29;10(1):12737. doi: 10.1038/s41598-020-69673-w. PMID 32728189
- [Background] Ranjan AK, Briyal S, Khandekar D, Gulati A. Sovateltide (IRL-1620) affects neuronal progenitors and prevents cerebral tissue damage after ischemic stroke. Can J Physiol Pharmacol. 2020 Sep;98(9):659-666. doi: 10.1139/cjpp-2020-0164. Epub 2020 Jun 23. PMID 32574518
- [Background] Gulati A, Hornick MG, Briyal S, Lavhale MS. A novel neuroregenerative approach using ET(B) receptor agonist, IRL-1620, to treat CNS disorders. Physiol Res. 2018 Jun 27;67(Suppl 1):S95-S113. doi: 10.33549/physiolres.933859. PMID 29947531
- [Background] Briyal S, Nguyen C, Leonard M, Gulati A. Stimulation of endothelin B receptors by IRL-1620 decreases the progression of Alzheimer's disease. Neuroscience. 2015 Aug 20;301:1-11. doi: 10.1016/j.neuroscience.2015.05.044. Epub 2015 May 27. PMID 26022359
- [Background] Leonard MG, Prazad P, Puppala B, Gulati A. Selective Endothelin-B Receptor Stimulation Increases Vascular Endothelial Growth Factor in the Rat Brain during Postnatal Development. Drug Res (Stuttg). 2015 Nov;65(11):607-13. doi: 10.1055/s-0034-1398688. Epub 2015 Mar 25. PMID 25806822
- [Background] Briyal S, Shepard C, Gulati A. Endothelin receptor type B agonist, IRL-1620, prevents beta amyloid (Abeta) induced oxidative stress and cognitive impairment in normal and diabetic rats. Pharmacol Biochem Behav. 2014 May;120:65-72. doi: 10.1016/j.pbb.2014.02.008. Epub 2014 Feb 20. PMID 24561065
- [Background] Leonard MG, Gulati A. Endothelin B receptor agonist, IRL-1620, enhances angiogenesis and neurogenesis following cerebral ischemia in rats. Brain Res. 2013 Aug 28;1528:28-41. doi: 10.1016/j.brainres.2013.07.002. Epub 2013 Jul 11. PMID 23850649
- [Background] Leonard MG, Briyal S, Gulati A. Endothelin B receptor agonist, IRL-1620, provides long-term neuroprotection in cerebral ischemia in rats. Brain Res. 2012 Jun 29;1464:14-23. doi: 10.1016/j.brainres.2012.05.005. Epub 2012 May 9. PMID 22580085
- [Background] Leonard MG, Briyal S, Gulati A. Endothelin B receptor agonist, IRL-1620, reduces neurological damage following permanent middle cerebral artery occlusion in rats. Brain Res. 2011 Oct 28;1420:48-58. doi: 10.1016/j.brainres.2011.08.075. Epub 2011 Sep 7. PMID 21959172
- [Background] Keam SJ. Sovateltide: First Approval. Drugs. 2023 Sep;83(13):1239-1244. doi: 10.1007/s40265-023-01922-4. PMID 37486545
- [Background] Briyal S, Ranjan AK, Gulati A. Oxidative stress: A target to treat Alzheimer's disease and stroke. Neurochem Int. 2023 May;165:105509. doi: 10.1016/j.neuint.2023.105509. Epub 2023 Mar 11. PMID 36907516